CLINICAL TRIAL: NCT04925440
Title: A Double-blind, Placebo-controlled, Randomised Study to Assess the Effects of Bifidobacterium Longum 1714® in a Population With Low Mood
Brief Title: The Effects of Bifidobacterium Longum 1714® in a Population With Low Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PrecisionBiotics Group Ltd. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-133
Record Dates: First submitted 2021-06-04; First posted 2021-06-14 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Low Mood; Depressive Symptoms
MeSH Terms: conditions — Consciousness Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Probiotic capsules. Participants will consume 2 capsules once a day for 8 weeks.
  Interventions: Dietary Supplement: Bifidobacterium longum 1714® strain
- Placebo (Placebo Comparator): Placebo capsules. Participants will consume 2 capsules once a day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum 1714® strain — Probiotic capsules containing 5 x 10^9 CFUs, corn-starch and magnesium stearate.
  Arms: Probiotic
Dietary Supplement: Placebo — Capsules containing corn-starch and magnesium stearate only.
  Arms: Placebo

SUMMARY:
A randomised, double-blind, placebo-controlled clinical trial to evaluate the effect of 8 weeks of supplementation with Bifidobacterium longum 1714® strain on Beck's Depression Inventory-II Score in adults who experience low mood.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group study, designed to assess the effectiveness & safety of Bifidobacterium longum 1714® strain in people with low mood. The 8-week intervention study will be conducted in 168 adults, aged ≥18 to ≤70 years, who experience low mood, and experience mild or moderate depression, according to the Beck's Depression Inventory II (Total score 14-28). The study will consist of 4 visits over a 10 week period commencing with a screening visit. The second visit will be the baseline (start of intervention - either active or placebo), followed by third (mid-intervention), fourth (end of treatment). Questionnaires will be administered from the first to the fifth visit and safety and research bloods will be collected at each visit throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to give written informed consent.
2. Male or female adults aged between ≥18 to ≤70 years.
3. Participants with a BMI between ≥18.5 and ≤29.9 kg/m2.
4. Meet the DSM-5 criteria for major depressive disorder (MDD) at screening (V0) and at baseline (V1).
5. BDI-II (Beck's Depression Inventory II) total score of 14-28 (mild [14-19] or moderate [20-28] depression) at screening (V0) and at baseline (V1).
6. Be willing to maintain stable dietary habits and physical activity levels throughout the study period.
7. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator.

Exclusion Criteria:

1. Participants who are at risk of suicide.
2. Recent use of dietary supplements, probiotics, or other fermented foods that contain live bacteria within last 4 weeks.
3. Participant who has been on antibiotics during the past 3 months.
4. Participant with a malignant disease or any concomitant end-state organ disease and/or laboratory abnormalities considered by Investigators to be risky or that could interfere with data collection.
5. Participant who has a significant physical illness (including IBS, does not include people with controlled hypertension or type II diabetes).
6. Participant who is severely immunocompromised (HIV positive, transplant patient, on anti-rejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year).
7. Significant psychiatric diagnosis (e.g., bipolar) other than depression.
8. Participants who are on anxiolytics, anti-depressants, antipsychotics, anticonvulsants, centrally acting corticosteroids, opioid pain relievers, hypnotics, and/or prescribed sleep medication/ herbals (e.g., valerian, St. John's Wort).
9. Participants with a current history of drug (including illicit drug) and /or alcohol abuse at the time of enrolment.
10. Participants who are pregnant (determined by urine pregnancy test for all individuals of childbearing potential at screening, regardless of contraceptive use or relationship status), breastfeeding, or wish to become pregnant during the study.
11. Participants who are suffering from post-natal depression.
12. Participants currently of childbearing potential, but not using an effective method of contraception, as outlined below:

    1. Complete abstinence from intercourse two weeks prior to administration of Investigational Product, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the Investigational Product in cases where participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
    2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
    3. Sexual partner(s) is/are exclusively female.
    4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm) or contraceptive pill. The participant must be using this method for at least 2 weeks prior to use of the Investigational Product and at least 1 week following the end of the study.
    5. Use of any non-hormonal intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1 % per year. The participant must have the device inserted at least 2 weeks prior to the first Screening Visit, throughout the study, and 2 weeks following the end of the study.
13. Known allergy to any of the components of the test product.
14. Participation in a clinical study with an Investigational Product within 60 days before screening or plans to participate in another study during the study period.
15. Participant has a history of non-compliance or in the opinion of physician deemed unsuitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms assessed by the Beck Depression Inventory (BDI-II) | Change from baseline compared to placebo, assessed over 8 weeks of supplement intake
  Severity of depression as measured by the BDI-II (range 0-63, with higher scores reflecting worse outcome)

SECONDARY OUTCOMES:
Change in depression severity category assessed by the Patient Health Questionnaire-9 (PHQ-9) | Change from baseline compared to placebo, assessed over 8 weeks of supplement intake
  Depression Severity category scores are as follows: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Change in fatigue assessed by the Visual Analogue Scale (VAS) for fatigue. | Change from baseline compared to placebo, assessed over 8 weeks of supplement intake
  The instrument possesses 18 items which has two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10). Each item is scored from 0-100 with higher scores indicating more fatigue or more energy.
Change in subjective sleep quality, assessed by Pittsburgh Sleep Quality Index global score | Change from baseline compared to placebo, assessed over 8 weeks of supplement intake
  Minimum score is 0, maximum score is 21. Higher scores indicate worse sleep quality.
Change in stress assessed by the by Cohen's Perceived Stress Scale (PSS) | Change from baseline compared to placebo, assessed over 8 weeks of supplement intake
  The PSS is a 14 item questionnaire with each item scored from 0-4. The total score ranges from 0-56 with a higher score indication more stress.
Change in quality of life assessed by the Short Form-36 | Change from baseline compared to placebo, assessed over 8 weeks of supplement intake
  The SF-36 is a self-administered questionnaire comprising 36-items measuring eight health domains: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.
Changes in depressive symptoms assessed by the Beck Depression Inventory (BDI-II) | Change from baseline compared to placebo, assessed at 4 weeks of supplement intake
  Severity of depression as measured by the BDI-II (range 0-63, with higher scores reflecting worse outcome)
Changes in mood category assessed by the Beck Depression Inventory (BDI-II) | Change from baseline compared to placebo, assessed at 4 weeks of supplement intake
  Severity of depression as measured by the BDI-II (range 0-63, with higher scores reflecting worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Dinan, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland